CLINICAL TRIAL: NCT02135133
Title: A Phase II Study of Idelalisib (GS1101, CAL101) + Ofatumumab in Previously Untreated Chronic Lymphocytic Leukemia (CLL) and Small Lymphocytic Leukemia (SLL)
Brief Title: A Study of Idelalisib (GS1101, CAL101) + Ofatumumab in Previously Untreated CLL/SLL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Gilead Sciences (Industry); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Jennifer R. Brown, MD, PhD, Sponsor Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-309
Record Dates: First submitted 2014-04-24; First posted 2014-05-09 (Estimated); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — idelalisib; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Idelalisib & Ofatumumab (Experimental): Idelalisib will be given orally continuously at 150 mg BID. On day 57, ofatumumab will begin with the 300 mg dose, given after idelalisib is taken. Ofatumumab will then be administered at 1000 mg weekly to complete 8 weeks (days 64, 71, 78, 85, 92, 99, 106) throughout Cycles 3 and 4. This will be followed by monthly ofatumumab on weeks 20, 24, 28, 32 to complete 4 additional cycles (5-8). The overall induction treatment period will then be 8 months, comprised of two months of single agent idelalisib followed by 6 months of ofatumumab with idelalisib. After the completion of the induction treatment, idelalisib will continue indefinitely in arbitrarily defined 28 day cycles in all participants who have not had excessive toxicity and do not have progressive disease.
  Interventions: Drug: Idelalisib; Drug: Ofatumumab

INTERVENTIONS:
Drug: Idelalisib — 150 mg BID Oral Daily
  Other Names: GS1101
Drug: Ofatumumab — Ofatumumab will then be administered at 1000 mg weekly to complete 8 weeks (days 64, 71, 78, 85, 92, 99, 106) throughout Cycles 3 and 4. This will be followed by monthly ofatumumab on weeks 20, 24, 28, 32 to complete 4 additional cycles (5-8).
  Other Names: Arzerra

SUMMARY:
This research study is evaluating a combination of drugs called Ofatumumab and Idelalisib as a possible treatment for Chronic Lymphocytic Leukemia (CLL) and Small Lymphocytic Leukemia (SLL).

The main purpose of this study is to examine the combination of the two drugs, Ofatumumab and Idelalisib, in participants who have been diagnosed with CLL/SLL and have not previously received treatment but do require treatment. The investigators hope to observe how participants' disease will be impacted by this treatment and whether they will benefit more from combining these drugs together rather than taking them separately. Both of these drugs have been used in treatment for CLL / SLL and information from those research studies suggests that these drugs may help patients with CLL/SLL.

Ofatumumab is an antibody engineered in the lab against CD20, a protein on the surface of CLL cells, which is expressed in CLL. An antibody is a molecule your body creates to identify foreign substances so that it can destroy them. Ofatumumab has been FDA approved for treatment of CLL/SLL that has relapsed or progressed on other therapies. Idelalisib is a drug that blocks one of the signals inside the cells that cause this type of cancer to grow and survive. The investigators hope that combining Ofatumumab with Idelalisib will stop the growth of disease.

In this research study, the investigators are evaluating the side effects of combining these two drugs, gathering information on the CLL/SLL disease process and how the study affects the patient's cells, as well as assessing the outcome of the disease. This combination of drugs has been previously tested, and appeared to be well tolerated.

DETAILED DESCRIPTION:
Before the research starts (screening): After signing the consent form, the participant will be asked to undergo some screening tests or procedures to find out if they are eligible to be in this research study. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that the participant does not take part in the research study. If the participant has had some of these tests or procedures recently, they may or may not have to be repeated.

* A medical history, which includes questions about the participant's health, current medications, and any allergies.
* Physical examination, which includes vital signs, height, weight, and disease assessment by the size of the participant's spleen, liver, and lymph nodes.
* Performance status, which evaluates how the participant is able to carry on with their usual activities.
* An assessment of the patient's tumor by CT (Computerized Tomography) scan, MRI or PET (Positron Emission Tomography) scans,
* Bone marrow aspirate and biopsy: A study tube (plastic cylinder container that contains biopsy material) will be drawn during this biopsy to further assess the participant's disease status.
* Blood tests, a maximum of 24 teaspoons will be collected.
* Urine test.
* A blood pregnancy test
* A Hepatitis B and C test, will require blood sample.

If these tests show that the participant is eligible to participate in the research study, then the participant will be begin will begin the study treatment. If you do not meet the eligibility criteria, the participant will not be able to participate in this research study.

Additional research procedures to be performed at the time of screening:

• Blood tests, including baseline tests so that the investigators can measure any additional effect of the study drug and disease status

After the screening procedures confirm that you are eligible to participate in the research study:

If you take part in this research study, the participant will be given a study drug-dosing diary for each treatment cycle. Each treatment cycle lasts 28 days. The diary will also include special instructions for taking the study drugs.

* Study Drugs: The participant will first be given Idelalisib daily for two cycles of 28 days each. Idelalisib will be given orally. Once the participant completes 2 cycles of Idelalisib, then the participant will start to receive a combination of Ofatumumab and Idelalisib. This regimen will continue weekly to complete 8 weeks (two more cycles). This will be followed by monthly Ofatumumab and Idelalisib to complete 4 additional cycles (eight total). The overall treatment period will therefore be 8 months, comprised of two months of Idelalisib followed by 6 months of Ofatumumab with Idelalisib. After completing the 8-month treatment, the participant will likely continue Idelalisib. Restaging with CT scans will happen after Cycle 2, 4, and a final restage will occur 2 months after the completion of Ofatumumab. There will be a tumor response assessment done during a physical exam after Cycle 8.
* Clinical Exams: During all cycles the participant will have a physical exam and will be asked questions about their general health and specific questions about any problems that they might be having and any medications they may be taking.
* Scans (or Imaging tests): The investigator will assess the participant's tumor by CT scan. Restaging with CT scans will happen after Cycle 2, 4, and a final restage will occur 2 months after the completion of Ofatumumab.
* Bone marrow aspirate and biopsy: will be conducted to see if the bone marrow has tumor cells. A study tube will be drawn during this biopsy to further assess the patient's disease status
* Blood tests

Additional Blood Tests:

Blood Tests will be performed throughout the study so that the Investigator can measure any additional effect of the study drug and disease status. These tests will be taken on the days listed below before the participant receive study drug, on some days additional blood will be drawn after they receive study drug.

Cycle 3 Day 1 Cycle 3 Day 8 Cycle 3 Day 15 Cycle 4 Day 21 (last weekly Ofatumumab dose) Cycle 5 Day 1 (first monthly Ofatumumab dose) Cycle 8 Day 1 (last monthly Ofatumumab dose) 2 months after Ofatumumab therapy completed 6 months after Ofatumumab therapy completed

Planned Follow-up:

Once the participant has completed the study treatment, the participant will be monitored until they start a new type of treatment or are removed from the study. During this time the participant will meet with your research physician every 3 or 6 months.

The investigator would like to keep track of the participant's medical condition for the rest of their life. The investigator would like to do this by calling the participant on the telephone once a year to see how the participant is doing. Keeping in touch with the participant and checking their condition every year helps the investigator look at the long-term effects of the research study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* Subjects must have CLL / SLL, as documented by a history at some point of an absolute peripheral blood B cell count > 5000, with a monoclonal B cell population co-expressing CD19, CD5, and CD23, or if CD23 negative, then documentation of the absence of t(11;14) or cyclin D1 overexpression. Alternatively patients with lymphadenopathy in the absence of circulating disease will also be eligible for this study if lymph node biopsy establishes the diagnosis of CLL with the above immunophenotype.
* Participants must have measurable disease (lymphocytosis > 5,000, or palpable or CT measurable lymphadenopathy > 1.5 cm, or bone marrow involvement >30%).
* Subjects must not have received any prior systemic therapy for CLL and currently have an indication for treatment as defined by the IWCLL 2008 Guidelines:
* Massive or progressive splenomegaly; OR
* Massive lymph nodes, nodal clusters, or progressive lymphadenopathy; OR
* Grade 2 or 3 fatigue; OR
* Fever ≥ 100.5°F or night sweats for greater than 2 weeks without documented infection; OR
* Presence of weight loss ≥ 10% over the preceding 6 months; OR
* Progressive lymphocytosis with an increase of ≥ 50% over a 2-month period or an anticipated doubling time of less than 6 months; OR
* Evidence of progressive marrow failure as manifested by the development of or worsening of anemia and or thrombocytopenia.
* ECOG performance status <2 (see Appendix A).
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of idelalisib or ofatumumab in participants <18 years of age, children are excluded from this study.
* Participants must have normal organ and marrow function as defined below:
* creatinine <2.0 times upper normal limit, total bilirubin <1.5 times upper normal limit (unless due to disease involvement of liver, hemolysis or a known history of Gilbert's disease)
* ALT <2.5 times upper normal limit (unless due to disease involvement of liver) alkaline phosphatase <2.5 times upper normal limit (unless due to disease involvement of the liver or bone marrow)
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Participants who have had any prior systemic therapy for CLL, or chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) for some other indication prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to ofatumumab or idelalisib.
* Subjects who have current active hepatic or biliary disease (with exception of participants with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 weeks prior to enrollment, whichever is longer, or currently participating in any other interventional clinical study
* Other past or current malignancy that could interfere with the interpretation of outcome. Subjects who have been free of active malignancy for at least 2 years, or have a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma, or whose malignancy will not interfere with the interpretation of study results, are eligible.
* Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active Hepatitis C.
* History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae
* Known HIV positive. HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with idelalisib. In addition, these individuals are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to randomization, congestive heart failure (NYHA III-IV), and arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities.
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the participant.
* Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HB DNA test will be performed and if positive the subject will be excluded.
* If HBV DNA is negative, subject may be included but must undergo HBV DNA PCR testing at least every 2 months from the start of treatment until 12 months post treatment. Prophylactic antiviral therapy may be initiated at the discretion of the investigator.
* Positive serology for hepatitis C (HC) defined as a positive test for HepC Ab, in which case reflexively perform an HC RIBA immunoblot assay or hepatitis C viral load to confirm the result. If the confirmatory test is negative the subject will be eligible.
* Pregnant or lactating women.
* Women of childbearing potential, including women whose last menstrual period was less than one year prior to screening, unable or unwilling to use adequate contraception from study start to 30 days after the last dose of protocol therapy. Adequate contraception is defined as hormonal birth control, intrauterine device, double barrier method or total abstinence.
* Male subjects unable or unwilling to use adequate contraception methods from study start to 30 days after the last dose of protocol therapy.
* Participants using concomitant corticosteroids are allowed as long as the subject is on the equivalent of 20mg/day or less of prednisone and has been on a stable dose for at least two weeks prior to initiating therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-06; Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Brown, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Lampson BL, Kim HT, Davids MS, Abramson JS, Freedman AS, Jacobson CA, Armand PA, Joyce RM, Arnason JE, Rassenti LZ, Kipps TJ, Fein J, Fernandes SM, Hanna JR, Fisher DC, Brown JR. Efficacy results of a phase 2 trial of first-line idelalisib plus ofatumumab in chronic lymphocytic leukemia. Blood Adv. 2019 Apr 9;3(7):1167-1174. doi: 10.1182/bloodadvances.2018030221. PMID 30967392
- [Derived] Lampson BL, Kasar SN, Matos TR, Morgan EA, Rassenti L, Davids MS, Fisher DC, Freedman AS, Jacobson CA, Armand P, Abramson JS, Arnason JE, Kipps TJ, Fein J, Fernandes S, Hanna J, Ritz J, Kim HT, Brown JR. Idelalisib given front-line for treatment of chronic lymphocytic leukemia causes frequent immune-mediated hepatotoxicity. Blood. 2016 Jul 14;128(2):195-203. doi: 10.1182/blood-2016-03-707133. Epub 2016 May 31. PMID 27247136

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients screened between 16 June 2014, and 14 March 2016, and 27 patients ultimately received at least 1 dose of study therapy
Period: Overall Study
Arm/Group | Idelalisib & Ofatumumab
Started | 27
Completed | 12
Not Completed | 15
Not completed — Adverse Event | 10
Not completed — regulatory mandate | 5

BASELINE CHARACTERISTICS:
Arm/Group | Idelalisib & Ofatumumab
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: years] | 69 [57 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Not of Hispanic Origin | 26
  Black/African American, not of Hispanic Origin | 1
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: The overall response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on IWCLL 2008 criteria.
Time Frame: Disease evaluated on Cycle 2 day 22 (Restage end of cycle 2), Cycle 10 day 1 (Final Restage 2 months after end of ofa therapy) and off treatment prior to cycle 10. Treatment duration is median 243 days with range of 9-620 days.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Idelalisib & Ofatumumab
Number analyzed (Participants) | 27
proportion of participants | 0.89 [0.77 to 1]

2. Secondary Outcome: Complete Response Rate (CRR)
Description: The overall response rate (ORR) was defined as the proportion of participants achieving CR based on IWCLL 2008 criteria.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Idelalisib & Ofatumumab
Number analyzed (Participants) | 27
proportion of participants | 0.037 [-0.03 to 0.11]

3. Secondary Outcome: Median Progression-Free Survival (PFS)
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration between randomization and documented disease progression (PD) or death, or is censored at time of last dsease assessment.
Time Frame: Disease evaluated on Cycle 2 day 22, Cycle 10 day 1 and off treatment prior to cycle 10. In long term, survival follow-up yearly. The median follow up time among survivors was 32.2 months (range 13, 35).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib & Ofatumumab
Number analyzed (Participants) | 27
months | NA [NA to NA] — Median and range not statistically reachable by Kaplan-Meier method because no enough events

ADVERSE EVENTS:
Time Frame: AEs were evaluated on treatment cycle 1-8 weekly, restage cycle 4 day 2, cycle 10 day 1, and off treatment prior to cycle 10. AE evaluation period is median 243 days with range of 9-620 days. Same with mortality.
Description: Serious adverse events (AEs) were defined as events with treatment-attribution of possibly, probably or definitely and grade 4 or higher per CTCAEv4. All remaining events regardless of treatment attribution were classified as Other AEs. Maximum grade toxicity by type for a patient over time was calculated. No further data is available to specify classification of other beyond the general term.
Arm/Group | Idelalisib & Ofatumumab
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 6/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib & Ofatumumab (N=27)
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 4
Neutrophil count decreased (Investigations) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib & Ofatumumab (N=27)
Alanine aminotransferase increased (Investigations) | 13
Aspartate aminotransferase increased (Investigations) | 13
Neutrophil count decreased (Investigations) | 11
Fever (General disorders) | 11
Diarrhea (Gastrointestinal disorders) | 10
Fatigue (General disorders) | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Nausea (Gastrointestinal disorders) | 7
Infusion related reaction (Injury, poisoning and procedural complications) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Chills (General disorders) | 4
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 4
General disorders and administration site conditions - Other, specify (General disorders) | 4
Anemia (Blood and lymphatic system disorders) | 3
Colitis (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dysgeusia (Nervous system disorders) | 3
Edema limbs (General disorders) | 3
Infections and infestations - Other, specify (General disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Alkaline phosphatase increased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 2
Blood bilirubin increased (Investigations) | 2
Bronchial infection (Infections and infestations) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Lung infection (Infections and infestations) | 2
Malaise (General disorders) | 2
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 2
Allergic reaction (Immune system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Esophageal pain (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Flu like symptoms (General disorders) | 1
Headache (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Lip infection (Infections and infestations) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Skin infection (Infections and infestations) | 1
Stomach pain (Gastrointestinal disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Upper respiratory infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT02135133/Prot_SAP_000.pdf